CLINICAL TRIAL: NCT04534660
Title: A Feasibility Study to Evaluate Preliminary Safety and Effectiveness of SMI-01 as a Tissue Filler
Brief Title: Preliminary Safety and Effectiveness of SMI-01 as a Tissue Filler
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sofregen Medical, Inc. (Industry)
Collaborators: Symbio, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SOF-001
Record Dates: First submitted 2020-07-10; First posted 2020-09-01 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Nasolabial Fold; Cheek Augmentation

STUDY DESIGN:
Intervention Model Description: This FDA approved feasibility study model includes 2 single groups, one for each indication (Cheek augmentation N=15; Nasolabial Fold Correction N=15). Both will receive the same treatment (SMI-01). Findings from the feasibility study will be used to inform study design for the Pivotal study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Nasolabial Fold (Experimental): SMI-01 is an injectable device comprising silk particles distributed in a hydrogel carrier. The intervention will be administed once, at the Day 1 visit. An optional touch-up treatment is allowed at the Day 30 visit.
  The study treatment facial areas are the Right and Left nasolabial fold. The Treating Investigator will inject SMI-01 into the mid to deep dermis for correction of moderate to severe wrinkle and folds. The Treating Investigator will determine the appropriate volume of SMI-01 to be injected during initial and touch-up treatment(s).
  Interventions: Device: SMI-01
- Cheek Augmentation (Experimental): SMI-01 is an injectable device comprising silk particles distributed in a hydrogel carrier. The intervention will be administed once, at the Day 1 visit. An optional touch-up treatment is allowed at the Day 30 visit.
  The midface constitutes the area of the face below the eyes and between the nose and the left or right ear. The study treatment facial areas are the Right and Left cheeks. The Treating Investigator will inject SMI-01 deeply (subcutaneous and/or supraperiosteal plane) for cheek augmentation to correct age-related volume deficiency in the midface, i.e., zygomaticomalar region, anteromedial cheek, and/or submalar region
  Interventions: Device: SMI-01

INTERVENTIONS:
Device: SMI-01 — SMI-01 is a device consisting of silk particles in a hydrogel carrier.

SUMMARY:
Multicenter (two clinical sites), unblinded, no control group, prospective feasibility study. Subject participation may last up to 24 months after enrollment. Treatment will be performed at Day 1 and optionally at Day 30, with the primary safety and effectiveness evaluation at 2 months. Subjects will continue extended follow-up evaluations at 4, 6, 12, 18 and 24 months after the final injection.

The duration and follow-up schedule will be identical, independent of treatment performed.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant, non-breastfeeding females, 22 to 65 years old.
2. Sign the Informed Consent form and the Authorization for Use and Release HIPAA form prior to any study-related procedures being performed.
3. Willing to comply with the requirements of the study, including sequential photography or imaging; willing to abstain from any plastic surgical or cosmetic procedures of the head or neck for the 24 months of the study (including but not limited to laser or chemical resurfacing, facelift, and other filler treatments).
4. Willing to avoid any intentional changes in weight, and avoid initiating any strict weight loss or weight gain programs.
5. Agrees to refrain from seeking other treatment for the treated condition during thestudy.
6. If the subject is a female of childbearing potential (sexually active and not sterile nor postmenopausal for at least 1 year), she must have a negative urine pregnancy test have used an acceptable contraception method for at least 30 days prior to enrollment, and agree to use an acceptable method of contraception for the duration of the study. The following are considered acceptable methods of birth control for the purpose of this study: oral contraceptives, contraceptive patches, contraceptive implant, vaginal contraceptive (NuvaRing®), double barrier methods (e.g., condom and spermicide), contraceptive injection (Depo-Provera®), intrauterine device (IUD), hormonal IUD (Mirena®), and abstinence with a documented second acceptable method of birth control if the subject becomes sexually active.

Inclusion Criteria Specific for Treatment Indications:

Cheek Augmentation:

8. Seeking augmentation therapy for the midface with a Midface Volume Scale (MFVS) score of a 1 (mild loss midface volume loss and or presence of mild concavity) or 2 (moderate midface volume loss and/or presence of moderate concavity) on each side of the face as assessed by the Treating Investigator.

9. Accept the obligation not to receive any other facial procedures or treatments affecting facial volume deficit at any time during the study.

Nasolabial Fold Correction:

10. Seeking augmentation therapy for the nasolabial folds with two fully visible nasolabial folds with Wrinkle Severity Rating Scale score of 3 or 4 (moderate or severe).

11. Accepts the obligation not to receive any other facial procedures or treatments affecting facial nasolabial fold deficit at any time during the study.

Exclusion Criteria:

1. Female subjects who are pregnant, breastfeeding, intending to become pregnant during the study, or who do not agree to use an acceptable form of birth control during the study.
2. Subjects who have a body mass index (BMI) of ≥ 30.
3. A history of allergy or hypersensitivity to injectable hyaluronic acid gel.
4. A history of allergy or hypersensitivity to silk.
5. Presentation on the face of any of the following: cysts, acne, rosacea, rashes or hives, infection, psoriasis, herpes zoster, actinic keratosis or any other disease that , in the opinion of the investigator, may result in changes in facial contour, edema of the face or otherwise interfere with study assessments.
6. Subjects who have undergone the following: 1) chemical peels, 2) microdermabrasion, 3) dermabrasion, or 4) needling procedures anywhere on the face or neck within 6 months prior to study treatment and throughout the study.
7. Subjects who received injectable neurotoxins on the face or neck area within 6 months prior to study treatment and throughout the study.
8. Subjects who have undergone facial treatment with a hyaluronic acid (HA) tissue filler within 12 months prior to study treatment and throughout the study.
9. Subjects who used deoxycholic acid treatment or other fat-reducing agents within 12 months prior to study treatment and throughout the study.
10. Subjects who have undergone mesotherapy, highintensity focused ultrasound (HIFU), high-intensity focused electromagnetic energy (HIFEM), or any other Energy Based Devices on the face within 12 months of the study and throughout the study. This also includes all intense pulsed light treatments, lasers (all), and RF treatments of any kind, photodynamic therapy, photomodulation with low level light sources (including laser light).
11. Subjects who have undergone facial treatment with a non-HA tissue filler (e.g., collagen, calcium hydroxylapatite, Poly-L-lactic Acid) within 18 months prior to study treatment and throughout the study.
12. Subjects who have ever undergone facial plastic surgery, tissue grafting, or received permanent facial implants (e.g., polymethyl methacrylate, polyacrylamide, silicone, fat transfer procedures or adipose matrix products, polytetrafluoroethylene, lifting threads, absorbable sutures) anywhere in the face or neck, or is planning to be implanted with any of these products during the course of the study.
13. Subjects who have severe malocclusion or dentofacial or maxillofacial deformities as judged by the Treating Investigator. Subjects planning to undergo extensive dental procedures such as dental implants, multiple tooth extractions, or oral surgery should not participate. Minor dental procedures such as teeth cleaning and repair of caries are not exclusionary.
14. Evidence of scar-related disease or delayed healing activity within the past 12 months.
15. Evidence of scar at the intended treatment region on the face.
16. History of keloid formation or hypertrophic scars.
17. History of bleeding disorders or connective tissue disorders or granulomatous diseases (sarcoidosis etc).
18. Presence of any wound or infection on the face.
19. Subjects with a midface volume deficit due to congenital defect, trauma, abnormalities in adipose tissue related to immune-mediated diseases such as generalized lipodystrophy (e.g., juvenile dermatomyositis), partial lipodystrophy (e.g., Barraquer-Simons syndrome), inherited disease, or HIV-related disease or HIV therapy.
20. The presence of any contraindication to the implant procedures in a relevant period before study entry (per the Treating investigator's judgment).
21. Subjects on the following therapy within 10 days of undergoing study device injections: a) prescribed anticoagulation therapy, thrombolytics, or inhibitors of platelet aggregation. Subjects are advised not to stop their prescribed therapy without consultation with their treating physician or primary care physician; b) nonsteroidal anti-inflammatory drugs (NSAIDs), or other substances known to increase coagulation time (e.g., herbal supplements with garlic or gingko, Vitamin E in excess of 50 IU per day). Subjects who will withhold such therapy for 10 days before AND after any injection session may participate.
22. Subjects on systemic (oral/injectable) corticosteroids or immunomodulatory/ immunosuppressive medications within 30 days prior to treatment. Subjects using topical steroids on the face within 14 days prior to treatment start and throughout the study.
23. Use of prescription wrinkle treatment (example: topical retinoids) or topical adapalene within 4 weeks (28 days) prior to treatment and throughout the study. Use of sunscreens and continued therapy with some cosmeceuticals (e.g., alpha hydroxyl acids, glycolic acids, or retinol-containing products) is allowed if the regimen was established ≥ 90 days prior to enrollment.
24. A history of severe allergies or multiple allergies manifested by anaphylaxis.
25. The presence of any condition that, in the opinion of the investigator, makes the subject unable to complete the study per protocol (e.g., subject not likely to avoid other facial cosmetic treatments).
26. Subjects not likely to stay in the study for up to 24 months because of other commitments, concomitant conditions, or past history.
27. Subjects with facial tattoo or facial hair that may interfere with diagnosis or evaluation of treatment.
28. The presence of known allergies, uncommon resistance, or hypersensitivity reactions to local topical anesthetics or nerve blocking agents (if such products are intended to be used for that subject).
29. History of or presence of cancerous or pre-cancerous lesions in the area to be treated.
30. Subjects who are immunocompromised or immunosuppressed.
31. Subjects who are employed by (or a relative of) the Treating Investigator, Site staff, Sponsor, or representative of the Sponsor.
32. Have received any investigational product within 30 days prior to study enrollment or be planning to participate in another investigation during the course of this study.
33. Subjects anticipated to be unreliable; or subjects who have a concomitant condition that might confuse or confound study treatments or assessments in the opinion of the investigator.
34. Subjects with "unattainable expectations."

    Exclusion Criteria Specific for Treatment Indication:

    Cheek Augmentation:
35. Subjects with an MFVS score of 0 (none to minimal midface volume loss with no apparent concavity) or 3 (severe midface volume loss and or severe concavity with apparent bony prominence) on the right or left midface as rated by the Treating Investigator.

    Nasolabial Fold Correction:
36. Subjects with a WSRS score of ≤ 2 (absent or mild) on the right or left nasolabial fold as rated by the Treating Investigator.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
To obtain clinician feedback on overall ease of use of device on a scale of 0 -10 (0 being not easy and 10 being most easy) | Initial Treatment, Day 1
  The Investigator will assess overall ease of use by the device by circling the appropriate number on the Numerical Rating Scale (NRS) from 0 being not easy to 10 being most easy.
Patient reported incidence of CTR's and any treatment emergent adverse events | Day 30
  Subject self-evaluation of Common treatment site responses (CTR's) and any treatment emergent adverse events as recorded in the Subject's 30-day diary. A diary will be dispensed to record CTR's responses such as erythema, tenderness, moderate swelling, pruritus or any allergic symptoms or possible systemic reaction such as a rash, arthralgia, myalgia that occurs at any time during the observation period.
Patient reported severity (mild, moderate or severe) of CTR's and any treatment emergent adverse events | Day 30
  Subject self-evaluation of Common treatment site responses (CTR's) and any treatment emergent adverse events as recorded in the Subject's 30-day diary. A diary will be dispensed to record CTR's responses such as erythema, tenderness, moderate swelling, pruritus or any allergic symptoms or possible systemic reaction such as a rash, arthralgia, myalgia that occurs at any time during the observation period.
Patient reported duration of CTR's and any treatment emergent adverse events | Day 30
  Subject self-evaluation of Common treatment site responses (CTR's) and any treatment emergent adverse events as recorded in the Subject's 30-day diary. A diary will be dispensed to record CTR's responses such as erythema, tenderness, moderate swelling, pruritus or any allergic symptoms or possible systemic reaction such as a rash, arthralgia, myalgia that occurs at any time during the observation period.
Investigator reported incidence of CTR's and any treatment-emergent adverse events | Month 2 after the last treatment
  The Treating Investigator will evaluate Common treatment site responses (CTR's) and any treatment emergent adverse events at the in-clinic visit.
Investigator reported duration of Common treatment site responses (CTR's) and any treatment-emergent adverse events | Month 2 after the last treatment
  The Treating Investigator will evaluate and document the subject's safety response to the Silk Restore treatment.
Investigator reported severity (mild, moderate or severe) of Common treatment site responses (CTR's) and any treatment-emergent adverse events | Month 2 after the last treatment
  The Treating Investigator will evaluate and document the subject's safety response to the Silk Restore treatment.
Change in midface volume retention measured by Sofregen's Midface Volume Scale (MFVS) for Cheek Augmentation subjects only | Month 2 after the last treatment
  Preliminary evaluation of the effectiveness of SMI-01 will be determined by the Treating Investigator's score of the subject's treatment using Sofregen's proprietary MFVS scale. The MFVS measures midface volume loss on a scale of 0 (none to minimal) to 3 (severe).
Change in wrinkle severity measured by Wrinkle Severity Rating Scale (WSRS) for Nasolabial fold correction subjects only | Month 2 after the last treatment
  Preliminary evaluation of the effectiveness of SMI-01 will be determined by the Treating Investigator's score of the subject's treatment using the WSRS. The WSRS measures wrinkle severity on a scale of 1 (absent) to 5 (extreme).

CONTACTS AND LOCATIONS:
Overall Officials: Leslie S. Baumann, MD, Principal Investigator — Baumann Cosmetic & Research Institute; Stacy Smith, MD, Principal Investigator — California Dermatology & Clinical Research Institute
Locations (2):
- United States (2):
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Baumann Cosmetic & Research Institute, Miami, Florida

IPD SHARING:
Plan to Share IPD: No